CLINICAL TRIAL: NCT02529072
Title: AVeRT: Anti-PD-1 Monoclonal Antibody (Nivolumab) in Combination With DC Vaccines for the Treatment of Recurrent Grade III and Grade IV Brain Tumors
Brief Title: Nivolumab With DC Vaccines for Recurrent Brain Tumors
Acronym: AVERT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gary Archer Ph.D. (Other)
Collaborators: Bristol-Myers Squibb (Industry); Duke Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Gary Archer Ph.D., Assistant Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00065241
Record Dates: First submitted 2015-08-12; First posted 2015-08-19 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Malignant Glioma; Astrocytoma; Glioblastoma
MeSH Terms: conditions — Glioma; Astrocytoma; Glioblastoma | interventions — Nivolumab; lentiviral minigene vaccine of COVID-19 coronavirus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Experimental): Patients will receive nivolumab 3 mg/kg IV every 2 weeks for 8 weeks followed by surgery. Following resection, nivolumab and DC vaccine will be administered every 2 weeks (± 1) for a total of 3 vaccines, followed by biweekly treatment with nivolumab and monthly DC vaccinations for a total of 5 more vaccines. Patients will continue to receive nivolumab every 2 weeks until progression.
  Interventions: Drug: nivolumab; Biological: DC
- Group II (Experimental): Patients will initially receive the fourth cycle of nivolumab then receive nivolumab 3 mg/kg IV and DC vaccine every 2 weeks for a total of 3 vaccines, and then surgery. Subsequent to surgery, the patient will resume biweekly treatment with nivolumab and monthly DC vaccinations for a total of 5 more vaccines. Patients will continue to receive nivolumab every 2 weeks until progression.
  Interventions: Drug: nivolumab; Biological: DC

INTERVENTIONS:
Drug: nivolumab — Nivolumab is a fully human monoclonal antibody that targets the programmed death-1 (PD-1) cluster of differentiation 279 cell surface membrane receptor. PD-1 is a negative regulatory molecule expressed by activated T and B lymphocytes. Binding of PD-1 to its ligands, programmed death-ligands 1 and 2, results in the down-regulation of lymphocyte activation. Inhibition of the interaction between PD-1 and its ligands promotes immune responses and antigen-specific T cell responses to both foreign antigens as well as self-antigens. Nivolumab is expressed in Chinese hamster ovary cells and is produced using standard mammalian cell cultivation and chromatographic purification technologies. The clinical study product is a sterile solution for parenteral administration.
  Other Names: BMS-936558; MDX1106
Biological: DC — DCs are potent immunostimulatory cells that continuously sample the antigenic environment of the host and specifically activate cluster of differentiation 4 positive (CD4+) and cluster of differentiation 8 positive (CD8+) T-cells and B-cells. They are at the crossroads of many of the elegant networks of the immune system, and DCs represent the most promising contemporary biologic entity for realizing the promise of immunotherapy. Potent immune responses and encouraging clinical results have been seen in Phase I and II human clinical trials in systemic cancers. Numerous animal studies and the investigator's institution's humans studies have demonstrated potent antitumor responses using DC-based immunotherapy against MGs.
  Other Names: DC vaccine; pp65 DC vaccine; Human CMV pp65-LAMP mRNA-pulsed autologous DCs; CMV pp65 DCs

SUMMARY:
Patients will be randomized to one of two treatment arms - Group I and Group II. Group I will receive nivolumab monotherapy until surgical resection, and Group II will receive nivolumab alone and with DC vaccine therapy until surgical resection. During surgical resection blood and tumor samples will be assessed and compared. Following surgery, both groups will continue to receive DC vaccines (total of 8) and nivolumab therapy until confirmed progression.

DETAILED DESCRIPTION:
This two-arm randomized trial will evaluate the safety of nivolumab in combination with DC vaccinations for the treatment of bevacizumab-naïve subjects with first or second recurrent, resectable World Health Organization (WHO) Grade III and IV malignant gliomas (MGs). Up to 66 patients will be enrolled and treated with the goal of accruing 30 patients (15 per arm) that will receive nivolumab and at least 3 vaccines. After enrollment, leukapheresis will be done for generation of DC vaccines and immunologic monitoring. All subjects will undergo standard of care tetanus booster vaccination with 0.5 mL of Td (tetanus and diphtheria toxoids adsorbed) intramuscularly (I.M.) into the deltoid muscle to ensure adequate immunity to the tetanus antigen. Subjects will initially return every 2 weeks and receive approximately 3 infusions of nivolumab 3 mg/kg IV while the DC vaccines are being prepared from the initial leukapheresis and will then be randomized 1:1 to one of 2 arms (Group I: nivolumab only pre-surgery; Group II: nivolumab with DC vaccines pre-surgery). Patients who are unable to tolerate nivolumab will be withdrawn from the study and replaced. Patients whose DCs or Peripheral Blood Lymphocytes (PBLs) fail to meet release criteria will continue to receive nivolumab only and will not undergo repeat leukapheresis. For patients whose leukapheresis yields less than 4 vaccines, a repeat leukapheresis may be obtained a minimum of 2 weeks from the previous leukapheresis (and may be repeated as needed) if stable. Peripheral blood will be drawn for immune monitoring prior to treatment with the 4th cycle of nivolumab (first post-randomization infusion of nivolumab).

Group I Treatment Plan (Nivolumab Only Pre-Surgery) After randomization, patients in Group I will receive nivolumab 3 mg/kg IV every 2 weeks x approximately 8 weeks. The subject will then undergo surgical resection of tumor within approximately 1-3 weeks. Approximately 2-4 weeks later, leukapheresis is repeated for generation of DC vaccines and immunologic monitoring. Approximately 1 day to 2 weeks after leukapheresis, the subject will resume nivolumab 3mg/kg IV every two weeks with DC vaccine administration intradermally (i.d.) for a total of 3 vaccines. At the time of the third DC vaccine, patients will receive vaccine site pre-conditioning. A single dose of Td toxoid (1 flocculation unit (Lf) in 0.4 milliliters (mL) of saline) will be administered to a single side of the groin i.d. (as described above for all vaccine administrations 12-24 hours prior to the third DC vaccine, which is always given bilaterally at the groin site. At the vaccine #3 visit, prior to vaccine # 3 administration, erythema and induration measurements will be taken of pre-conditioning site. Group I subjects will then receive monthly DC vaccine administrations intradermally for 5 months or until progression (whichever comes first).Total vaccines to be administered will be 8 post-surgery unless subject is removed. Nivolumab will continue until progression. At the clinic visit following the last vaccine (#8), subjects will have peripheral blood drawn for immune monitoring prior to infusion of nivolumab.

Group II Treatment Plan (Nivolumab with DC Vaccines Pre-Surgery) After randomization, patients in Group II will receive the fourth cycle of nivolumab then receive nivolumab 3 mg/kg IV along with DC vaccines intradermally every 2 weeks x approximately 6 weeks for a total of 3 vaccines. At the time of the third DC vaccine, patients will receive vaccine site pre-conditioning. A single dose of Td toxoid (1 Lf in 0.4 mL of saline) will be administered to a single side of the groin i.d. 12-24 hours before the third DC vaccine, which is always given bilaterally at the groin site. At the vaccine #3 visit, prior to vaccine #3 administration, erythema and induration measurements will be taken of pre-conditioning site.The subject will then undergo surgical resection of tumor within approximately 1-3 weeks. Approximately 2-4 weeks later, leukapheresis is repeated for generation of DC vaccines and immunologic monitoring. Approximately 1 day to 2 weeks after leukapheresis, the subject will resume nivolumab 3mg/kg IV every two weeks. When DC vaccines have completed processing and are available for administration, monthly DC vaccine administrations as described above will be administered for 5 months or until progression (whichever comes first). Total vaccines to be administered will be 8 (3 pre- and 5 post-surgery) unless subject is removed. Nivolumab will continue until progression. At the clinic visit following the last vaccine (#8), subjects will have peripheral blood drawn for immune monitoring prior to infusion of nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years of age
* First or second recurrence of MG (WHO Grade III or IV glioma or astrocytoma) in surgically accessible areas with prior histologic diagnosis of MG
* Bevacizumab-naïve - no prior exposure to Bevacizumab
* Karnofsky Performance Status (KPS) of ≥ 70%
* Radiation Therapy (RT) with ≥ 45 Gray (Gy) tumor dose, completed ≥ 8 weeks prior to study entry
* Laboratory values must meet the following criteria:

  1. White Blood Count (WBC) ≥ 2000/microliters (uL)
  2. Neutrophils ≥ 1500/uL
  3. Platelets ≥ 100x103/uL
  4. Hemoglobin ≥ 9.0 g/dL
  5. Serum creatinine ≤ 1.5x the upper limit of normal (ULN) or creatinine clearance (CrCl)≥ 40 mL/min (using the Cockcroft-Gault formula) c. Female CrCl = (140 - age in years) x weight in kg x 0.85 /72 x serum creatinine in mg/dL d. Male CrCl = (140 - age in years) x weight in kg x 1.00/72 x serum creatinine in mg/dL
  6. Aspartate Aminotransferase (AST) ≤ 3x ULN
  7. Alanine Aminotransferase (ALT) ≤ 3x ULN
  8. Bilirubin≤ 1.5x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
  9. Subjects must have resting baseline O2 saturation by pulse oximetry of ≥ 92% at rest.
* Patients of child bearing potential or with partners of child-bearing potential must practice recommended contraceptive methods to prevent pregnancy during treatment and for 5 months after the last dose of nivolumab for women, 7 months after the last dose of nivolumab for men, and for 6 months after the last dose of bevacizumab for subjects receiving bevacizumab.

Exclusion Criteria:

* Contrast-enhancing tumor component crossing the midline, multi-focal tumor, or tumor dissemination (subependymal or leptomeningeal)
* Clinically significant increased intracranial pressure (e.g., impending herniation), uncontrolled seizures, or requirement for immediate palliative treatment
* Pregnant or need to breast feed during the study period (Negative human chorionic gonadotropin (β-HCG) test required), or unable to maintain use of contraception while on study and for 31 weeks after the last dose of nivolumab
* Active infection requiring treatment or an unexplained febrile (> 101.5o F) illness
* Known immunosuppressive disease, autoimmune disease or human immunodeficiency virus infection, Hepatitis B or Hepatitis C
* Known allergy or hypersensitivity to tetanus, or any other tetanus or diphtheria toxoid-containing vaccine, or any component of this vaccine (i.e., aluminum phosphate, formaldehyde)
* Known severe (Grade 3 or 4) infusion-related allergy or hypersensitivity to any monoclonal antibody
* Previous radiation therapy with anything other than standard radiation therapy (such as previous stereotactic radiosurgery) or previous treatment with an immune checkpoint inhibitor (i.e., nivolumab, pembrolizumab, ipilimumab)
* Unstable or severe intercurrent medical conditions such as severe heart (New York Association Class 3 or 4) or lung (FEV1 < 50%) disease, uncontrolled diabetes mellitus
* Corticosteroid use > 4 mg/day at time of consent
* Prior inguinal lymph node dissection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Peters, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I | Group II
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I | Group II | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (6.6) | 61.2 (1.8) | 57.1 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Safety of Administering DC Vaccines With Nivolumab
Description: The percentage of patients who experience unacceptable toxicity during combination treatment by arm is tabulated. Unacceptable toxicity is defined as any grade 3, 4, or 5 adverse event that is possibly, probably, or definitely related to either nivolumab or DC vaccination treatment during concurrent treatment, or any Grade 2 drug-related uveitis or eye pain or blurred vision that does not respond to topical therapy and does not improve to Grade 1 severity within the re-treatment period OR requires systemic treatment. In addition, any complication following resection (ex. excessive intracranial bleeding, delays in wound healing) that are prolonged longer than 4-6 weeks post-surgery will be considered an unacceptable toxicity.
Time Frame: 12 months
Population: All randomized patients are included in this analysis
Measure: Number; unit: Percentage of patients
Arm/Group | Group I | Group II
Number analyzed (Participants) | 3 | 3
Percentage of patients | 0 | 0

2. Secondary Outcome: Overall Survival
Description: Survival is defined as the time between first initiation of nivolumab and death, or last follow-up if the patient remains alive. The Kaplan-Meier estimator will be used to describe the overall survival (OS) experience of all patients. Median OS is presented. Patients who are not able to tolerate nivolumab and are removed from the study will not be included in these analyses. Patients for whom DC vaccines cannot be manufactured will not be included in the survival analyses.
Time Frame: approximately 4 years from study initiation
Population: All randomized patients are included in this analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group I | Group II
Number analyzed (Participants) | 3 | 3
months | 8.0 [5.7 to 8.3] | 15.3 [4.73 to NA] — The upper limit is not estimable due an insufficient number of patients and events

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time between treatment initiation and initial progression or death, or date of last follow-up if the patient remains alive without disease progression. The Kaplan-Meier estimator will be used to describe the PFS experience of all patients. Median PFS is presented. Patients who are not able to tolerate nivolumab and are removed from the study will not be included in these analyses. Patients for whom DC vaccines cannot be manufactured will not be included in the survival analyses. Tumor assessment will be made using Response Assessment in Neuro-Oncology (RANO) criteria, which defines progressive disease as an increase by at least 25% in the sum of the products of perpendicular diameters from the baseline scan, a significant increase in T2/FLAIR non-enhancing lesions, or clinical decline
Time Frame: 6 to 48 months from study initiation
Population: All randomized patients are included in this analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group I | Group II
Number analyzed (Participants) | 3 | 3
months | 4.3 [2.1 to 5.3] | 6.3 [4.7 to 10.7]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Group I | Group II
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I (N=3) | Group II (N=3)
Meningitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1
Injury, poisoning and procedural complications - Other, Specify: L EAR LACERATION (Injury, poisoning and procedural complications) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I (N=3) | Group II (N=3)
Anemia (Blood and lymphatic system disorders) | 2 | 3
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Endocrine disorders - Other, Specify: ELEVATED TSH; POSSIBLY RELATED TO NIVO (Endocrine disorders) | 0 | 1
Blurred vision (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, Specify: POLYDIPSIA (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Edema face (General disorders) | 0 | 1
Edema limbs (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Gait disturbance (General disorders) | 1 | 0
Pain (General disorders) | 1 | 2
Infections and infestations - Other, Specify: HEAD INCISION IRRITATION (Infections and infestations) | 0 | 1
Infections and infestations - Other, Specify: SMALL CUT ON L HAND (Infections and infestations) | 1 | 0
Infections and infestations - Other, Specify: YEAST INFECTION (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal and connective tissue disorders - Other, Specify: STEROID MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify: SWOLLEN NECK (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dysphasia (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 1 | 1
Memory impairment (Nervous system disorders) | 1 | 1
Nervous system disorders - Other, Specify: FACIAL DROOP (Nervous system disorders) | 0 | 1
Nervous system disorders - Other, Specify: WEAKNESS IN R HAND (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, Specify: COLD (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, Specify: CLAMMY AND COOL SKIN (Skin and subcutaneous tissue disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT02529072/Prot_SAP_000.pdf